Investigating the Use of Temporary Abstinence and Expressive Writing for Reducing Problematic Gaming

23 September 2024

# PARTICIPANT INFORMATION SHEET & CONSENT FORM



NUS-IRB Reference Code: NUS-IRB-2023-1037

1. Protocol title

Gaming Routine, Writing, and Online Gaming

2. Principal Investigator and co-investigator(s), if any, with the contact number and organization:

Principal Investigator: Dr. Ryan Hong, PhD

Organization: Department of Psychology, NUS

Telephone Number:

Co-Investigator: Mr. Jonathan Tan

Organization: Department of Psychology, NUS

Telephone Number:

3. What is the purpose of this research?

You are invited to participate in a research study that examines the relationship between gaming routine, writing, and online gaming behaviour. This information sheet provides you with information about the research study. Please read the information below and ask questions about anything you don't understand before deciding whether or not to take part.

4. Who can participate in the research? What is the expected duration of my participation? What is the duration of this research?

Singapore citizens or Permanent Residents between 18 and 35 years old, who are able to read and write English proficiently and are non-professional regular online gamers willing to temporarily take a break from gaming for 7 consecutive days. Online games refer to video games that are played over the Internet using computers, smartphones, tablets, or gaming consoles (e.g., PlayStation, Xbox, Nintendo switch). These do not include offline games (e.g., arcade machines, board/card games, offline video games) or secondary games that are part of a primarily non-gaming application (e.g., mini games in e-commerce applications like Shopee or Lazada).

You will be required to attend a short Zoom briefing (approximately 15 minutes), respond to 1 initial survey (approximately 1 hour), follow a prescribed gaming routine and engage in 4 writing exercises (1 every alternate day, approximately 15 minutes each) for one week, respond to 1 post-survey one week later (approximately 30 minutes), and 1 follow-up survey 1 month later (approximately 45 minutes). The estimated total time commitment for attending the briefing and completing all surveys and exercises is 3 - 3.5 hours.

- 5. What is the approximate number of research participants involved? The research team intends to recruit 450 participants for this study.
- 6. What will be done if I take part in this research study?

You will be required to first attend a short online briefing via Zoom where a member of the research team will share more details about the procedures and to answer any questions about the study. After the briefing, you will complete an initial online survey in one sitting on the same day. Before the end of the day, you will receive an email with information about the prescribed gaming routine that you will need to follow for 7 consecutive days. You will also be asked to complete a writing exercise on your daily experiences once every alternate day during that same week. You will complete 4 such writing exercises and are required to submit them before the end of that day. Please note that the research team is unable to provide you with a replacement writing exercise if you miss the deadline for submission, and your participation in the research may be automatically terminated if you fail to complete at least 3 out of 4 writing exercises during the designated days. After 1 week has ended, you will be asked to complete a post survey in one sitting. Lastly, one month after completion of the post survey, you will also be asked to complete a final follow-up online survey in one sitting. All survey links and reminders will be sent to your email address. The research team may also reach out to you using the mobile phone number you provided for scheduling the briefing session and sending reminders to complete the surveys.

Please take each question seriously and carefully, as the time and effort you spend on each question in the surveys will affect our evaluation of the quality of your answer. Please note that the research team may either request you to reattempt the survey or automatically terminate your participation in the research if your response fails a basic quality check.

Some research designs require that the full extent of the study not be explained prior to participation. Although we have described the general nature of the tasks that you will be asked to perform, the full intent of the study will not be explained to you until after the completion of the study. At that time, we will provide you with a full debriefing which will include an explanation of the hypothesis that was tested and other relevant background information pertaining to the study. You will also be given an opportunity to ask any questions you have about the hypothesis and the procedures used in the study.

# 7. How will my privacy and the confidentiality of my research records be protected?

Only members of the NUS research team will have access to your identifiable information (e.g., email address, contact information). Identifiable information will never be used in a publication or presentation. All identifiable information and research data will be coded (i.e. only identified with a code number) at the earliest possible stage of the research. Identifiable information will be discarded upon the completion of the research. Quotes from your responses in the surveys and writing exercises may be used in research outputs anonymously, subject to your consent.

All data collected will be kept in accordance with the University's Research Data Management Policy. Research data used in any publication will be kept for a minimum of 10 years before being discarded. All personal data will be destroyed after all study-related administration (e.g., reimbursement) are completed.

#### 8. What are the possible discomforts and risks for participants?

This study is of minimal risk, yet participants may experience discomfort when answering the survey or engaging in the writing exercises. If you experience any

discomfort with respect to some of the questions being asked in the survey, you are free to take breaks or stop your participation at any time. Similarly, if you feel that you are "flipping out" or losing control when writing about your daily experiences in the writing exercises, you can simply proceed to write about another topic.

#### 9. What is the compensation for any injury?

No injury and thus no compensation is expected. However, if you follow the directions of the PI in charge of this research study and you are injured, the NUS will pay the medical expenses for the treatment of that injury. By giving your consent, you will not waive any of your legal rights or release the parties involved in this study from liability for negligence.

#### 10. Will there be reimbursement for participation?

You will be reimbursed a total of \$120 for your time and effort in adhering to the study requirements and completion of all surveys and exercises; attending the Zoom briefing, completing the initial survey, following your prescribed gaming routine for 1 week, completing the 4 writing exercises according to the writing instructions, and completing the post survey and 1-month follow-up survey. If not all surveys are completed, reimbursement will be pro-rated. Participants will be reimbursed based on which surveys or exercises are completed: (a) attending the Zoom briefing and completion of the initial survey will lead to a reimbursement of \$20, (b) completion of each writing exercise according to the writing instructions will lead to a reimbursement of \$5 each, with a bonus \$7 for the completion of all 4 writing exercises, (c) completion of the post survey will lead to a reimbursement of \$8, (d) completion of the 1-month follow-up survey will lead to a reimbursement of \$25, and (e) a bonus of \$40 for your time and effort for adhering to our entire research protocol and completing all required surveys (i.e., following your prescribed gaming routine, submitting at least 3 out of 4 valid writing exercises, as well as responses for all surveys passing our basic quality check).

If you choose to withdraw midway through the initial survey or 1-month follow-up survey, you will be reimbursed \$10 for the initial survey or \$12.50 for the 1-month follow-up survey if you completed at least half of the questionnaire battery.

If your response fails a basic quality check, your participation in the research may be terminated automatically, and you will not be reimbursed for the survey that fails the check. Reimbursement will not be provided if we discovered that you have participated more than once or if you are not a Singapore citizen/PR, even if you proceed to complete all the surveys and exercises. Please also note that attending the Zoom briefing is a strict requirement for participating in this study. Likewise, no reimbursement will be provided If you do not attend the Zoom briefing, even if you proceed to complete all the surveys and exercises in the research.

### 11. What are the possible benefits to me and to others?

There is no direct benefit to you by participating in this research study. The knowledge gained may benefit the public in the future through the understanding of the relationship between gaming routine, writing and online gaming behaviour over time.

### 12. Can I refuse to participate in this research?

Yes, you can. Your decision to participate in this research study is voluntary and completely up to you. You can also withdraw from the research at any time without giving any reasons, up to 1 week of completing the final follow-up survey, by informing the Principal Investigator or Co-Investigator and all your data collected will be discarded. This is because the research team will not be able to trace which data belong to you once the personal data are discarded and no longer linked to your responses.

#### 13. Whom should I call if I have any questions or problems?

Please contact the Co-Investigator, Mr. Jonathan Tan at <email>, for all research-related matters and in the event of research-related injuries.

For an independent opinion specifically regarding the rights and welfare of research participants, you may contact a staff member of the National University of Singapore Institutional Review Board at telephone (+65) 6516 1234 [Mondays to Thursdays from 8.30am to 6pm, and Fridays from 8.30am to 5.30pm, except public holidays] or email at irb@nus.edu.sg.

Version No. 3, dated 23rd Sep 2024

## **Consent Form**

#### **Protocol title:**

Gaming Routine, Writing, and Online Gaming

#### Principal Investigator with the contact number and organization:

Principal Investigator: Dr. Ryan Hong, PhD

Organization: Department of Psychology, NUS

Telephone Number:

I hereby acknowledge that:

1. I have agreed to take part in the above research.

- 2. I have read a copy of this information sheet that explains the use of my data in this research. I understand its contents and agree to donate my data for the use of this research.
- 3. I can withdraw from the research at any point of time from the start of the study and up to 1 week of completing my participation in the study, by informing the Principal Investigator or Co-Investigator and all my data will be discarded.
- 4. I will not have any financial benefits that result from the commercial development of this research.
- 5. I agree / do not agree\* to the use of quotes from my responses to the surveys and writing exercises in research outputs anonymously. I understand that no identifiable information will be linked to the quotes used in any research outputs.

If you consent to participate in this study, please click on the "I consent" option, and continue.

If you do not consent to participate in this study, please click on the "I do not consent" option.